CLINICAL TRIAL: NCT03530241
Title: Sensitivity and Specificity of Fluorescent Cholangiography to Detect Bile Duct Stones in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Fluorescent Cholangiography and Bile Duct Stones
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Lars Lang Lehrskov, MD, Hvidovre University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IFC4
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Gall Stones, Common Bile Duct
Keywords: fluorescence; cholangiography; cholecystectomy, laparoscopic
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRCP positive (Experimental)
  Interventions: Diagnostic Test: Presence of bile duct stones
- MRCP negative (Active Comparator)
  Interventions: Diagnostic Test: Non-presence of bile duct stones

INTERVENTIONS:
Diagnostic Test: Presence of bile duct stones — MRCP verified gall stones in the bile ducts
  Arms: MRCP positive
Diagnostic Test: Non-presence of bile duct stones — MRCP without bile duct stones
  Arms: MRCP negative

SUMMARY:
Background. X-ray cholangiography has a high sensitivity and specificity of detecting bile duct stones and is the gold standard. There are no studies describing the sensitivity and specificity of IFC for bile duct stone detection.

Research question. What is the sensitivity of IFC to visualize bile duct stones? Method. Prospective study with 40 patients undergoing planned laparoscopic cholecystectomy with preoperative magnetic resonance cholangiopancreatography (MRCP) (gold standard) and intraoperative IFC, X-ray cholangiography and choledochuscopy in that order.

Primary outcome. Sensitivity of visualization of bile duct stone by fluorescent cholangiography and secondary outcome is visualization of anatomy.

ELIGIBILITY:
Inclusion criteria

* Patients suspected of having bile duct stones by either blood samples, MRCP or medical history (see definitions)
* Patient age ≥ 18 years
* Preoperative MRCP
* Operation performed by a project surgeon

Exclusion criteria

* Open cholecystectomy (including conversion from laparoscopic to open)
* Acute cholecytitis or cholangitis
* Pancreatitis
* Iodine or indocyanine green allergy
* Liver or renal insufficiency
* Thyrotoxicosis
* Cholecystectomy not the primary surgical procedure
* Pregnancy or lactation
* Legally incompetent for any reason
* Withdrawal of inclusion consent at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity | 120mins
  Sensitivity and specificity of visualization of bile duct stones by intraoperative fluorescent cholangiography

SECONDARY OUTCOMES:
Visualization | 120mins
  Visualization of the extrahepatic bile ducts

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Lehrskov, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Holte, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided